CLINICAL TRIAL: NCT05520983
Title: BEhavioral Health Stratified Treatment (BEST) to Optimize Transition to Adulthood for Youth With Intellectual and/or Developmental Disabilities (IDD)
Brief Title: BEhavioral Health Stratified Treatment (BEST) Study for Youth With Intellectual and/or Developmental Disabilities (IDD)
Acronym: BEST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Wellesley College (Other); The Arc of Illinois (Unknown); University of Chicago (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Benjamin Van Voorhees, MD, MPH, Professor and Head, Department of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CHAIRb 21092401
Record Dates: First submitted 2022-06-28; First posted 2022-08-30 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Depression; Anxiety; Transition
Keywords: Youth; Intellectual and developmental disabilities; Care coordination; Transition to adulthood; Cognitive-behavioral therapy; Adolescents; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Developmental Disabilities | interventions — Therapeutics; Caregivers

STUDY DESIGN:
Intervention Model Description: Comparative-effectiveness study of two different care coordination models
Who Masked: Outcomes Assessor
Masking Description: Assessors at Wellesley Centers for Women B.E.S.T. Call Center (BCC) will be blinded to conditions and the assessment measures that they complete do not involve collecting any measures of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Illinois MCHB Care Coordination (Active Comparator): MCHB Care Coordination is funded through the Social Security Act of 1935 Title V Maternal and Child Health Services Block Grant Program, this is the oldest and most universal care coordination model for children with I/DD. The University of Illinois Chicago Division of Specialized Care for Children (DSCC) is the Illinois (IL) state Title V MCHB care coordination agency and has annual contact with over 19,000 families and youth in IL. MCHB (known as DSCC) Care Coordination involves: comprehensive needs assessments, person-centered planning, and linkage to health care and social resources. MCHB care coordination has established efficacy, feasibility, and acceptability in improving child and family functioning, youth health, and health care access.
  Interventions: Other: Maternal Child Health Bureau (MCHB) Care Coordination
- Illinois MCHB Care Coordination + CHECK tiered behavioral health (Experimental): MCHB Care Coordination plus CHECK: includes all elements of MCHB care coordination, described above, plus the CHECK program. The CHECK program consists of a trained, behavioral health care team; an evidence-based treatment algorithm to classify risk for depression and anxiety (minimal, subclinical and clinical symptomatology) and guide treatment advancement [Tier 1/selective: cognitive behavioral psycho-education; Tier 2/indicated: cognitive-behavioral prevention groups; Tier 3/treatment: individualized or group cognitive-behavioral treatment (CBT)]; as well as structures and processes to support communication, coordination and data sharing between MCHB care coordinators and CHECK staff.
  Interventions: Behavioral: Adapted Teens Achieving Mastery over Stress (TEAMS) Treatment; Behavioral: Adapted Teens Achieving Mastery over Stress (TEAMS) Prevention; Behavioral: Adapted Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT); Other: Strengthening Families; Other: Virtual psycho-educational discussion groups for caregivers and participants; Other: Maternal Child Health Bureau (MCHB) Care Coordination

INTERVENTIONS:
Behavioral: Adapted Teens Achieving Mastery over Stress (TEAMS) Treatment — Teens Achieving Mastery over Stress (TEAMS) has been adapted for use with youth with I/DD. The intervention consists of virtual, manualized treatment groups for 10 weekly, 75-minute sessions plus 6 monthly, 60-minute sessions. Caregivers of participants will meet twice: weeks one and 16.
  Arms: Illinois MCHB Care Coordination + CHECK tiered behavioral health
Behavioral: Adapted Teens Achieving Mastery over Stress (TEAMS) Prevention — Teens Achieving Mastery over Stress (TEAMS) has been adapted for youth with I/DD. TEAMS Prevention is a 10-session group depression prevention program teaching teens how to deal with stress and negative moods, and ways to manage low mood based on cognitive behavioral therapy (CBT) principles and strategies. Efficacy has been demonstrated by several trials over time.
  Arms: Illinois MCHB Care Coordination + CHECK tiered behavioral health
Behavioral: Adapted Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT) — Competent Adulthood Transition with Cognitive-behavioral & Interpersonal Training (CATCH-IT) has been adapted for youth with I/DD. CATCH-IT is an internet-based depression prevention program that targets decreasing modifiable risk factors while enhancing protective factors in at-risk adolescents, and that includes a parent program. It has been shown to be safe, feasible, and efficacious. All adolescents will receive 8 engagement texts during their participation in the study - at 1-week, 1-month, 6-weeks, and 2-, 3-, 5-, and 5.5-months - to encourage participation in the online modules.
  Arms: Illinois MCHB Care Coordination + CHECK tiered behavioral health
Other: Strengthening Families — The Strengthening Families caregiving curriculum is an evidence-based, self-directed, virtual skills training for caregivers. Information and instructions on accessing the Strengthening Families parenting skills training curriculum will be included on the virtual resource website https://strengtheningfamilieslessons.org/.
  Arms: Illinois MCHB Care Coordination + CHECK tiered behavioral health
Other: Virtual psycho-educational discussion groups for caregivers and participants — The BEST project will host a total of 10 virtual psycho-educational workshops per year (5 for participants and 5 for caregivers) for the duration of the intervention period of the study. Workshops will be delivered remotely via Zoom and facilitated by graduate students in health/behavioral health. Simultaneous language interpreter services will be provided. Principles of universal design in learning will be applied to the content and delivery of workshops. Workshops are an optional resource available to all participants and families in the intervention condition. Topics for the virtual discussion groups will be determined based on pilot data and input from participants and caregivers.
  Arms: Illinois MCHB Care Coordination + CHECK tiered behavioral health
Other: Maternal Child Health Bureau (MCHB) Care Coordination — MCHB Care Coordination, funded through the Social Security Act of 1935 Title V Maternal and Child Health Services Block Grant Program, is the oldest and most universal care coordination model for children with I/DD. MCHB Care Coordination involves: comprehensive needs assessments, person-centered planning, and linkage to health care and social resources. MCHB care coordination has established efficacy, feasibility, and acceptability in improving child and family functioning, youth health, and health care access.

SUMMARY:
Many youth with disabilities and their families receive "care coordination services" from a state Maternal and Child Health Bureau (MCHB) agency. MCHB care coordination services help youth with disabilities get the medical care and social services they need to be healthy. Complex HEalth Care for Kids (CHECK) developed a program to combine mental health treatment and care coordination services for youth with disabilities. The goal of this study is to see whether a care coordination program that treats depression and anxiety (MCHB care coordination + CHECK) is better than a care coordination program (MCHB care coordination alone) that refers youth to mental health services in terms of making youth feel healthier, happier, and able to handle future challenges. The project team will test which care coordination approach is better at making youth with disabilities: (Aim 1) less anxious and depressed; (Aim 2) feel healthier, function better, and practice healthy habits; (Aim 3) improve their ability to manage their health. This study will also evaluate which approach makes (Aim 4) youth, caregivers, and providers feel more satisfied with their care coordination experience. This study will give youth with disabilities and their families information about what kinds of care coordination models are available, and better suited to their needs. The study team will reach out to 780 youth with intellectual and/or developmental disabilities, age 13-20 years old, who receive care coordination services from the state of Illinois MCHB. If these youth are eligible and agree to be in the study, they will be placed, by chance, into either MCHB care coordination alone or into the MCHB care coordination + CHECK program. In both groups, youth will have a care coordinator who helps them identify and make plans to meet their needs and provides referrals to services/resources. Youth in the MCHB care coordination + CHECK care coordination will get mental health treatment directly from CHECK staff if they report symptoms of depression or anxiety. Treatment may include an online program or group meetings that teach youth how to cope with negative thoughts and feelings. Youth in each group will be followed for 24 months and will receive gift cards for participating. Youth will be asked questions about anxiety and depression, health, functioning, ability to manage their health care, self-efficacy, and their experience with care coordination.

DETAILED DESCRIPTION:
Background and Significance : Youth (13-20 years) with intellectual and/or developmental disabilities (I/DD) often struggle with depression and anxiety disorders, which adversely impacts transition to adulthood. Integrated behavioral health care coordination, in which care coordinators and behavioral health specialists work together to provide systematic, cost-effective, patient-centered care, is an effective strategy to improve access to behavioral health services and address factors that impact transition to adulthood, including depression/anxiety symptoms. Current widely used care coordination models, such as Title V Maternal and Child Health Bureau (MCHB) care coordination (operating in > 40 states), do not include behavioral health services. Coordination of CarE for Complex Kids (CHECK), is a behavioral health risk classification and intervention delivery program that was designed for integration into care coordination programs, such as MCHB care coordination, and implemented under Centers for Medicare and Medicaid (CMS) Healthcare Innovation Award (#C1C1CMS331342-01-00; 2014-2018, $19.4 million, >6,000 youth enrolled). It is unknown whether an integrated behavioral health care coordination strategy, such as MCHB care coordination plus CHECK, would be more acceptable and lead to better youth health and transition outcomes, in comparison to standard care coordination (e.g., MCHB care coordination). Results would guide future investment in improving outcomes for youth with I/DD.

Aims: This study is a two-arm randomized clinical trial to evaluate the comparable efficacy of (1) MCHB Care Coordination alone vs. (2) MCHB Care Coordination plus CHECK in: (Aim 1) decreasing symptoms and episodes of depression and anxiety over time among at-risk transition-age youth with I/DD; (Aim 2) improving health behaviors, adaptive functioning and health related quality of life among transition-age youth with I/DD; (Aim 3) increasing health care transition (HCT) readiness among transition-age youth with I/DD; and (Aim 4) improving engagement and satisfaction with care coordination among stakeholders across multiple levels.

Comparators: 1. IL MCHB Care Coordination 2. IL MCHB Care Coordination + CHECK

1. MCHB Care Coordination: funded through the Social Security Act of 1935 Title V Maternal and Child Health Services Block Grant Program, this is the oldest and most universal care coordination model for children with I/DD. The University of Illinois at Chicago (UIC) Division of Specialized Care for Children (DSCC) is the Illinois (IL) state Title V MCHB care coordination agency and has annual contact with over 19,000 families and youth in IL. MCHB (known as DSCC) Care Coordination involves: comprehensive needs assessments, person-centered planning, and linkage to health care and social resources. MCHB care coordination has established efficacy, feasibility, and acceptability in improving child and family functioning, youth health, and health care access.
2. MCHB Care Coordination plus CHECK: includes all elements of MCHB care coordination, described above, plus the CHECK program. CHECK consists of: a trained, behavioral health care team; an evidence-based treatment algorithm to classify risk for depression and anxiety (minimal, subclinical and clinical symptomatology) and guide treatment advancement [Tier 1/selective: cognitive behavioral psychoeducation; Tier 2/indicated: cognitive-behavioral prevention groups; Tier 3/treatment: individualized or group cognitive behavioral treatment (CBT)]; as well as structures and processes to support communication, coordination and data sharing between MCHB care coordinators and CHECK staff. The CHECK Tiers are based upon the Coping with Depression-Youth curriculum and employ a psychoeducational approach to teach youth cognitive behavioral skills to prevent or reduce depression and anxiety symptoms and episodes (Clarke et al; integrative CBT model). The CHECK program was implemented within a large, community-based care coordination system, reached Level 6 integration (Full Collaboration in a Transformed /Merged Integrated Practice), and demonstrated feasibility, acceptability and favorable impacts on health, engagement and other outcomes.

Study Population: The investigators will recruit N=780 (N1=390; N2=390) transition-age youth with I/DD (13-20 years) from the IL MCHB Care Coordination program (i.e., DSCC), which serves a large racially, geographically, and socioeconomically diverse population across IL (23.65% Hispanic/Latino; 20.13% African American; 3.53% Asian; 50.20% White; 0.12% American Indian/Native Alaskan; 0.06% Native Hawaiian/other Pacific Islander) (57.00% male; 40.20% female; 2.70% transgender/non binary). Eligibility criteria include being a current DSCC participant, aged 13-20 years, with a minimum 4th grade reading level, and prior diagnosed I/DD. I/DD are chronic conditions, beginning at birth or prior to age 22 years, and include physical, learning, language, and/or behavioral impairments. Participants must be competent to consent. Exclusion criteria include severe intellectual disability (ID) (i.e., IQ<50) and reading below a 4th grade level. Assuming 10% loss to follow-up, the investigators require N = 780 for the 2-arm study.

Analytic Plan: The experimental design of the study is a 2 Group (MCHB care coordination vs. MCHB care coordination + CHECK intervention), 4 Times (0 baseline, 6, 12, and 24 months) repeated measures design. The goal is to determine whether the combination of MCHB care coordination plus CHECK yields greater improvement in patient outcomes over time than MCHB care coordination alone. The outcomes are continuous approximately normal multi-item scales (AIM 1: depression/anxiety symptomatology; AIM 2: health behaviors, adaptive functioning and health related quality of life; AIM 3: health care transition readiness; and AIM 4: engagement and satisfaction) which will be analyzed using linear mixed models (LMMs) that are the modern standard for analysis of repeated measures. The generalized linear mixed model (GLMM) will be used to analyze repeated outcomes that are categorical or counts (AIM 1: depression and anxiety episodes). In this design, contrasts can be used to test omnibus and group-specific (interaction) changes from baseline. Our primary model will include covariates for stratification variables (Z, W). Moreover, by introducing patient subgroups (S), it is possible to examine 3-way interactions (G T S) to test for the heterogeneity of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

A) Youth ages 13 through 20 years, B) who have an I/DD (caregiver/self-report), and C) are enrolled in MCHB care through the IL DSCC

Exclusion Criteria:

A) Participant has a severe ID (IQ <50) (caregiver/self-report); ( B) Participant has a reading/comprehension level below 4th grade (caregiver/self-report); or C) Participant is unable to consent to participate in the study based on the MacArthur Competency Assessment Tool Checklist of Questions (MacCAT-CR).

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 780 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptomatology | Baseline through 24 months
  The Patient Health Questionnaire Youths (PHQ-A) is a 9-item self-report measure of depressive symptomatology that has been shown to be both valid and reliable (α=.86-.89) (4-point Likert scale, 0-27 score range, higher score indicating more depressive symptoms/severity).This instrument has been used to assess depression in individuals with Autism Spectrum Disorder (ASD), cystic fibrosis and other I/DD.
Depressive Symptomatology (additional measures for those participating in Tiers 2 and 3) | Baseline through 24 months
  The Patient Health Questionnaire 8 (PHQ-8) is an 8-item self-report measure of depressive symptomatology that has been shown to be both valid and reliable (4-point Likert scale, 0-24 score range, higher score indicating more depressive symptoms/severity). This instrument is a version of the PHQ-9 that does not include a question regarding suicidality. Participants in Group B, Tier 2 will receive this instrument during the course of the Tier 2 intervention (online group sessions). Participants in Group B, Tier 3 will receive this instrument during the course of the Tier 3 intervention (online group sessions).
Anxiety Symptomatology | Baseline through 24 months
  The Generalized Anxiety Disorder (GAD-7) is a 7-item measure of anxiety symptomatology (4-point Likert scale, 0-21 score range, higher score indicating greater anxiety severity) that has been shown to be both valid and reliable (α=.92) and has been used to assess anxiety in individuals with ASD and other I/DD. Additionally, participants in Group B, Tier 2 will receive this instrument during the course of the Tier 2 intervention (online group sessions). Participants in Group B, Tier 3 will receive this instrument during the course of the Tier 3 intervention (online group sessions).
Major Depression Disorder and Anxiety Disorder | Baseline through 24 months
  The Mini-International Neuropsychiatric Interview for Children and Youths (MINI Kid) is a structured diagnostic interview for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) and International Classification of Diseases, Tenth Revision (ICD-10) psychiatric disorders in children and adolescents. The 72-item (yes/no response choices) sub-scales to identify depression and anxiety disorders will be utilized. These scales have been found to be both valid and reliable, and have been used with individuals with ASD and other I/DD.
Depressive Symptomatology of Caregiver | Baseline through 24 months
  The Patient Health Questionnaire (PHQ-9) is a 9-item adult-report measure of depressive symptomatology (4-point Likert scale, 0-27 score range, higher score indicating more depressive symptoms/severity) that has shown to be valid and reliable (α=.86-.89).
Anxiety Symptomatology of Caregiver | Baseline through 24 months
  The Generalized Anxiety Disorder (GAD-7) is a 7-item measure of anxiety symptomatology (4-point Likert scale, 0-21 score range, higher score indicating greater anxiety severity) that has been shown to be both valid and reliable (α=.92).

SECONDARY OUTCOMES:
Caregiver-Reported Adaptive Functioning | Baseline through 24 months
  The Waisman Activities of Daily Living (W-ADL) Scale is a 17-item caregiver-report survey of activities of daily living (3-point Likert scale, 0-34 score range, higher score indicating greater independence), specifically developed for adolescents/adults with I/DD. It has good criterion and construct validity.
Youth-Reported Adaptive Functioning | Baseline through 24 months
  The Waisman Activities of Daily Living (W-ADL) Scale is a 17-item self-report survey of activities of daily living (3-point Likert scale, 0-34 score range, higher score indicating greater independence), specifically developed for adolescents/adults with I/DD. It has good criterion and construct validity.
Health Related Quality of Life | Baseline through 24 months
  The Short Form 8 (SF-8) is an 8-item measure of health-related quality of life (5- or 6-point Likert scale) that has been used in population health and outcome studies. A higher standardized total score indicates better health. The instrument has high validity and test-retest reliability.
Health Behaviors - Risk Behaviors | Baseline through 24 months
  The Youth Risk Behavior Survey (YRBS) examines 6 areas of health-related behaviors among youth and young adults. Seven items related to physical activity (score range 0 to 7 days/week), screen time (score range <1hr to 5+ hours/day), and sleep (<4hr to 10+ hr/day) will be utilized. Higher scores indicate more physical activity each week, greater screen time each day, and more sleep each night. This survey has been found to be valid and reliable for diverse populations, including I/DD).
Health Behaviors - Substance Abuse | Baseline through 24 months
  The Car, Relax, Alone, Forget, Friends, Trouble (CRAFFT) screening tool is a 10-item (yes/no responses, with more yes responses indicating a higher probability of substance us/dependence), validated substance abuse screening tool for adolescents aged 12-21 years that is recommended by the American Academy of Pediatrics for preventive care screenings.
Transition Readiness of Youth and Caregivers | Baseline through 24 months
  The Transition Readiness Assessment Questionnaire (TRAQ) is a 20-item (5-point Likert scale, 20-100 score range, higher score indicating greater skill in areas important for transition to adult health care), valid and reliable (α=0.93) tool that captures self-management, self-advocacy, and health care utilization skills. The tool has been used with diverse youth with IDD. The instrument will be delivered to both participants and caregivers at baseline and 12 and 24-months.
Transition Readiness of Youth | Baseline through 24 months
  The Rotterdam Transition Profile (RTP) is a 6-item tool to summarize the transition profile of adolescents and young adults (3 or 4-point Likert scale, higher score indicating greater transition readiness), developed for use with individual with Cerebral Palsy.
Self-Efficacy | Baseline through 24 months
  The Generalized Self-Efficacy Scale (GSE) is a 10-item, valid and reliable (α=.76-.90) tool that captures the perceived ability to cope with adversity and perform various acts of daily living after experiencing a stressful life event (4-point Likert scale, 10-40 score range, higher score indicating greater self-efficacy). The instrument has been used with individuals with disabilities.
Integration of Care | At 12 months
  The Patient Assessment of Chronic Illness Care (PACIC) is a 20-item, self-report instrument (5-point Likert scale, 1-5 score range) with good internal reliability (α=0.93) and predictive validity that measures patient perceptions of care including delivery system follow-up and coordination. The instrument has 5 subscales (1-5 score range), and higher scores indicate better perceptions of care. The instrument has been used with individuals with I/DD. The instrument will be delivered to participants at 12-months.
Resilience | Baseline through 24 months
  The Connor Davidson-Resilience Scale (CD-RISC-10) is a 10-item, self-report instrument measuring resilience in terms of coping skills, including hardiness and persistence (4 levels of response, 0-40 score range, higher score indicating better coping skills). The instrument has good psychometric properties and has been used with individuals with I/DD, including ASD (α=.85).
Coping | Baseline through 24 months
  The Brief Coping Orientation to Problems Experienced (COPE) is a 28-item tool that measures 14 types of coping strategies using a 4-point Likert scale. The internal consistency of the 14 two-item sub-scales ranges from .49 (venting) to .98 (substance use). Sub-scale total scores range from 4-8, and higher scores indicate greater endorsement of the coping strategy. In a sample of youth seeking medical care, 13 of the 14 sub-scales had an internal consistency above. This instrument is used with individuals with chronic disabilities.
Perceived Stress of Youth and Caregivers | Baseline through 24 months
  The National Institutes of Health (NIH) Toolbox Perceived Stress is a 10-item, valid and reliable (α=.89-.91) instrument that measures subjective experience of stress (5-point Likert scale, 10-50 score range, higher score indicating greater perceived stress). The instrument has versions for those aged 13-17 years and those aged 18+ years. It has been used with individuals with neurological disorders.
Cognitive Style | Baseline through 24 months
  The Children's Cognitive Style Questionnaire (CCSQ) is a 30-item, valid and reliable instrument that measures negative cognitive style which makes individuals vulnerable to anxiety and depression (5-point Likert scale, 0-150 score range, higher score indicating greater negativity of cognitive style). The instrument has been used with both children and adults with disabilities.
Social Health - Peer Relationships | Baseline through 24 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Peer Relationships v2.0 is a 15-item valid and reliable instrument that measures relationships and social support (5-point Likert scale, 15-75 score range, higher score indicating stronger peer relationships). The instrument has been used with individuals with chronic disease and disability.
Stigma | Baseline through 24 months
  The Perceived Stigma in Intellectual and Developmental Disabilities Scale is a 10-item (yes/no, 0-10 score range, higher scores indicating greater perceived stigma) instrument with good reliability (.83) that measures the scope of stigma experiences across life domains. The instrument will be delivered to participants at baseline and 12 and 24-months.
Social Support of Caregiver | Baseline through 24 months
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item instrument with good validity and reliability (α=.94) that measures perceived social support from family, friends, and a significant other (7-point Likert scale, 7-84 score range, higher score indicating greater perceived social support). The instrument has been used with caregivers of children with I/DD.
Adverse Childhood Experiences | At 12 months.
  The Adverse Family Experiences (AFE) questionnaire was developed for the National Survey of Child Health. It was validated by a technical panel and has been used in numerous peer-reviewed studies, in which clinically meaningful associations between cumulative AFE scores and child health outcomes were demonstrated. The Adverse Family Experiences questionnaire consists of 9 questions (2-point Likert scale, 0-9 score range, higher score indicating AFEs) about children's exposure to the following: neighborhood violence, racial/ethnic discrimination, income hardship, caregiver divorce, incarceration, death, domestic violence, substance abuse, and mental illness. This instrument has been used with caregivers of individuals with I/DD. The instrument will be delivered to caregivers at 12-months.
Intervention Usability | At 12 months
  The Usefulness, Satisfaction, and Ease of Use Questionnaire (USE) is a 30-item, reliable (α =.97) measure of usability of technology and websites (30 items, self-report, 7-point Likert scale, 30-210 score range, higher score indicates greater usefulness, satisfaction, and ease of use). The instrument will be included for participants and caregivers at the end of the Tier 1 intervention (online module).
Intervention Acceptability | Baseline through 24 months
  The Acceptability of Intervention Measure (AIM) is a 4-item, self-report measure of implementation success that has strong psychometric properties and reliability (α=.89) (5-point Likert scale, 1-5 score range, higher score indicates greater acceptability of intervention). This instrument will be included for participants at the end of the Tier 2 and Tier 3 interventions (i.e., at the completion of the online group sessions). Participants and caregivers will report on the instrument at baseline, 12- and 24-months.
Health Behaviors - Law Enforcement Interaction | Baseline through 24 months
  The Personal Interests and Activities Subscale of the National Longitudinal Transition Study 2: Young Adult Questionnaire (NLTS2) includes 2-items (self-report, yes/no, yes indicates interaction with law enforcement) about youth interaction with law enforcement. The instrument will be delivered to participants at baseline and 12 and 24-months.

OTHER OUTCOMES:
Sociodemographic Information | Baseline through 24 months
  Participants will report on their date of birth, race/ethnicity, gender identity, household information, and school and employment status. They will also report on key demographics for the caregiver(s) they live with. Caregivers will also report on household/family information, including caregiver demographics, household structure, and socioeconomic status and insurance. They will also report on participant school and employment status. These items will be reported on at baseline and 24-months. Participants and caregivers will also report on the participant's clinical medication use and medical and psychiatric diagnoses at baseline, 12, and 24-months. At baseline, 12, and 24-months, participants and caregivers will also report on if the participant has ever (or currently) received individual or group therapy for mood or anxiety and if the participant has ever been hospitalized for depression or other mental health issues.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Berg, PhD, Principal Investigator — University of Illinois at Chicago; Benjamin W Van Voorhees, MD, MPH, Principal Investigator — University of Illinois at Chicago; Iulia Mihaila, PhD, Study Director — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Division of Specialized Care for Children, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White PH, Cooley WC; TRANSITIONS CLINICAL REPORT AUTHORING GROUP; AMERICAN ACADEMY OF PEDIATRICS; AMERICAN ACADEMY OF FAMILY PHYSICIANS; AMERICAN COLLEGE OF PHYSICIANS. Supporting the Health Care Transition From Adolescence to Adulthood in the Medical Home. Pediatrics. 2018 Nov;142(5):e20182587. doi: 10.1542/peds.2018-2587. Epub 2018 Oct 22. PMID 30348754
- [Background] Schwartz LA, Tuchman LK, Hobbie WL, Ginsberg JP. A social-ecological model of readiness for transition to adult-oriented care for adolescents and young adults with chronic health conditions. Child Care Health Dev. 2011 Nov;37(6):883-95. doi: 10.1111/j.1365-2214.2011.01282.x. PMID 22007989
- [Background] Jensen PT, Paul GV, LaCount S, Peng J, Spencer CH, Higgins GC, Boyle B, Kamboj M, Smallwood C, Ardoin SP. Assessment of transition readiness in adolescents and young adults with chronic health conditions. Pediatr Rheumatol Online J. 2017 Sep 9;15(1):70. doi: 10.1186/s12969-017-0197-6. PMID 28888223
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Johnson JG, Harris ES, Spitzer RL, Williams JB. The patient health questionnaire for adolescents: validation of an instrument for the assessment of mental disorders among adolescent primary care patients. J Adolesc Health. 2002 Mar;30(3):196-204. doi: 10.1016/s1054-139x(01)00333-0. PMID 11869927
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sheehan DV, Sheehan KH, Shytle RD, Janavs J, Bannon Y, Rogers JE, Milo KM, Stock SL, Wilkinson B. Reliability and validity of the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). J Clin Psychiatry. 2010 Mar;71(3):313-26. doi: 10.4088/JCP.09m05305whi. PMID 20331933
- [Background] Maenner MJ, Smith LE, Hong J, Makuch R, Greenberg JS, Mailick MR. Evaluation of an activities of daily living scale for adolescents and adults with developmental disabilities. Disabil Health J. 2013 Jan;6(1):8-17. doi: 10.1016/j.dhjo.2012.08.005. Epub 2012 Oct 17. PMID 23260606
- [Background] Fougeyrollas P, Noreau L, Bergeron H, Cloutier R, Dion SA, St-Michel G. Social consequences of long term impairments and disabilities: conceptual approach and assessment of handicap. Int J Rehabil Res. 1998 Jun;21(2):127-41. doi: 10.1097/00004356-199806000-00002. PMID 9924676
- [Background] Knight JR, Shrier LA, Bravender TD, Farrell M, Vander Bilt J, Shaffer HJ. A new brief screen for adolescent substance abuse. Arch Pediatr Adolesc Med. 1999 Jun;153(6):591-6. doi: 10.1001/archpedi.153.6.591. PMID 10357299
- [Background] Yiengprugsawan V, Kelly M, Tawatsupa B. SF-8TM Health Survey. Springer Netherlands; 2014:5940-5942.
- [Background] CDC. Youth Risk Behavior Survey: data summary and trends report, 2007-2017. Atlanta, GA: US Department of Health and Human Services, CDC; 2018. https://www.cdc.gov/healthyyouth/data/yrbs/pdf/trendsreport.pdf
- [Background] Donkervoort M, Wiegerink DJ, van Meeteren J, Stam HJ, Roebroeck ME; Transition Research Group South West Netherlands. Transition to adulthood: validation of the Rotterdam Transition Profile for young adults with cerebral palsy and normal intelligence. Dev Med Child Neurol. 2009 Jan;51(1):53-62. doi: 10.1111/j.1469-8749.2008.03115.x. Epub 2008 Nov 20. PMID 19021680
- [Background] Schwarzer R, & Jerusalem M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Lund AM. Measuring usability with the use questionnaire12. Usability interface. 2001;8(2):3-6.
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Schmittdiel J, Mosen DM, Glasgow RE, Hibbard J, Remmers C, Bellows J. Patient Assessment of Chronic Illness Care (PACIC) and improved patient-centered outcomes for chronic conditions. J Gen Intern Med. 2008 Jan;23(1):77-80. doi: 10.1007/s11606-007-0452-5. Epub 2007 Nov 21. PMID 18030539
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Background] Kupst MJ, Butt Z, Stoney CM, Griffith JW, Salsman JM, Folkman S, Cella D. Assessment of stress and self-efficacy for the NIH Toolbox for Neurological and Behavioral Function. Anxiety Stress Coping. 2015;28(5):531-44. doi: 10.1080/10615806.2014.994204. Epub 2015 Feb 10. PMID 25577948
- [Background] Abela JR. The hopelessness theory of depression: a test of the diathesis-stress and causal mediation components in third and seventh grade children. J Abnorm Child Psychol. 2001 Jun;29(3):241-54. doi: 10.1023/a:1010333815728. PMID 11411786
- [Background] Dewalt DA, Thissen D, Stucky BD, Langer MM, Morgan Dewitt E, Irwin DE, Lai JS, Yeatts KB, Gross HE, Taylor O, Varni JW. PROMIS Pediatric Peer Relationships Scale: development of a peer relationships item bank as part of social health measurement. Health Psychol. 2013 Oct;32(10):1093-103. doi: 10.1037/a0032670. Epub 2013 Jun 17. PMID 23772887
- [Background] Stuart H, Milev R, Koller M. The Inventory of Stigmatizing Experiences: Its development and reliability. World Psychiatry. 2005;4:35-39.
- [Background] Zimet GD, Dahlem NW, Zimet SG, Farley GK. The Multidimensional Scale of Perceived Social Support. Journal of Personality Assessment. 1988/03/01 1988;52(1):30-41. doi:10.1207/s15327752jpa5201_2
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Ali A, Strydom A, Hassiotis A, Williams R, King M. A measure of perceived stigma in people with intellectual disability. Br J Psychiatry. 2008 Nov;193(5):410-5. doi: 10.1192/bjp.bp.107.045823. PMID 18978324